CLINICAL TRIAL: NCT06483659
Title: Intravenous Oxytocin for Post Operative Pain After Minimally Invasive Hysterectomy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, John J. Kowalczyk, MD, Director of Fellowship Research, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024P001376
Record Dates: First submitted 2024-06-23; First posted 2024-07-03 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Oxytocin; Saline Solution

STUDY DESIGN:
Intervention Model Description: 152 study subjects who are having minimally invasive abdominal hysterectomy will be randomized into one of two treatment groups, the first group will receive Oxytocin I.V. infusion and the second group will receive Saline infusion, and both groups will be followed up with surveys for up to 3 months after surgery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization of the study medication will be performed by the investigational drug pharmacy and the unblinded key will be stored in a secure location in the pharmacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medication (Active Comparator): one group will receive Oxytocin infusion: 30 IU in 500 ml of 0.9% normal saline .
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): one group will receive 500 ml of 0.9% normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Intravenous Oxytocin infusion
  Other Names: Pitocin
  Arms: Medication
Drug: Placebo — 0.9% Saline
  Other Names: Normal Saline; 0.9% Saline
  Arms: Placebo

SUMMARY:
This is a randomized, double-blinded, placebo-controlled trial to compare the effectiveness of IV oxytocin infusion to placebo on peri-operative opioid consumption and reducing post-operative pain following a minimally invasive hysterectomy under general anesthesia.

DETAILED DESCRIPTION:
152 women will be randomized into one of two arms; participants in the first arm (Intervention) will receive oxytocin infusion, 30 IU in 500 ml IV infusion at a rate of 5 IU/h (83.33 ml/h), the second arm (Control) will receive 0.9% normal saline 500 ml IV infusion at the same rate of 83.3 ml/h. The primary care team (anesthesia, surgery, and nursing), the research team, and the patient will all be blinded to the research arm.

The investigational research pharmacy will perform randomization; participants will be randomized in a 1:1 ratio to receive either Oxytocin or Placebo (0.9% normal saline). Randomization will be blinded to investigators to prevent bias and ensure balance in treatment arms throughout the study. Participants, surgeons, clinicians, and raters will be blinded with respect to treatment assignments. The investigational pharmacy will prepare the study drug based on the randomization assignment received.

The investigators will identify patients who have been scheduled for an elective, minimally invasive hysterectomy at Brigham and Women's Hospital by reviewing the operating room booking schedule.

Patients will be pre-screened for inclusion and exclusion criteria. Subsequently, they will be recruited for participation in this study by phone/ MGB Zoom and will be consented by electronic consent.

Once the patient is recruited and consented, they will be randomized for either the intervention group (oxytocin IV infusion) or the control group (0.9% normal saline IV infusion).

An email will be sent to those who consent with a link to the secure REDCap system containing a set of baseline questionnaires to assess relevant medical and surgical history, pre-operative pain, analgesic medication use, and psychosocial variables.

Both groups (intervention and control) will be treated pre-operatively with the following Early Recovery After Surgery (ERAS) medications, as per usual institutional practice:

* acetaminophen 1,000 mg orally
* celecoxib 400 mg orally The Investigational Research Pharmacy will be informed and prepare blinded infusions for perioperative administration (oxytocin or placebo).

The primary anesthesiology team will receive either the study medication or placebo in a 500 ml bag labeled as "Oxytocin Study Drug for IV infusion".

A recommended "Intra-Operative Analgesia Management" algorithm will be given to the primary anesthetic team. The recommended algorithm for intra-operative analgesia management will include the following:

* Fentanyl 100 mcg IV for induction.
* Dexamethasone 8 mg IV after induction but prior to skin incision.
* Small, titrated doses of Hydromorphone IV boluses (0.2-0.4 mg) during the operation and before emergence, according to primary team judgment.
* Ketorolac 30 mg IV prior to skin closure, unless otherwise contraindicated.
* Avoidance of other multimodal analgesic agents not included in this protocol to limit confounders.

The infusion will be started after the skin incision and will continue until the infusion is completed or the post-anesthesia care unit (PACU) criteria are met, whichever occurs first.

Other aspects of each patient's routine clinical care will continue as per standard care at the attending physician's discretion under whom the patient is admitted, regardless of treatment arm status.

In the PACU, a brief postoperative pain questionnaire will be performed, including the Surgical Pain Scales (SPS).

The SPS is a validated scale consisting of 4 items that measure pain at rest, during normal activities, and during work/exercise and quantify the unpleasantness of worst pain. This scale has been validated in a number of different types of postoperative pain, including women after gynecologic surgery.

Vital signs, numeric rating scale (NRS) pain scores, and opioid consumption in PACU will be collected from the patient's medical record.

Patients whose surgery was converted to open, estimated blood loss (EBL) >500 ml, or any other surgical complication that necessitates hospitalization will be excluded from the trial.

For secondary outcomes, including total opioid consumption in 24, 48, and 72 hours and pain scores at postoperative day (POD)1, 2, and 3, an online survey will be done at POD1, 2, and 3, and follow-up will continue until 3 months post-op.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65 years old
* ASA category 1-3
* Scheduled to undergo minimally invasive hysterectomy
* No documented allergy to oxytocin

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) group 4 or greater
* Age >65 years old
* Additional surgical procedures including but not limited to minor laparotomy, omentectomy, cystectomy, vaginectomy, and/or ablation of endometriosis.
* Active opioid prescription of the equivalent of oxycodone >10 mg /day
* Opioid use disorder, including patients in treatment receiving naltrexone or Suboxone (Buprenorphine-naloxone)
* Allergies to any study medication: acetaminophen, celecoxib, ketorolac, fentanyl, hydromorphone, or oxycodone.
* Epidural/Regional anesthesia for intra-operative or post-operative pain.
* Inability to understand the questionnaires
* Intra-operative and post-operative exclusion: Procedure converted to open or extension of primary surgery, Intra-operative EBL >500 ml., Placement of epidural catheter or regional anesthesia at PACU for pain management, Hospitalization of the patient due to surgical or anesthetic complications

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | Between 2-4 hours after surgery completion (in the PACU)
  Assess the impact of a perioperative infusion of oxytocin on postoperative pain, the average patient pain scores measured as a mean Brief Pain Inventory in PACU after laparoscopic hysterectomy in treated and untreated groups will be compared

SECONDARY OUTCOMES:
Perioperative opioid consumption | From start of infusion until approximately 6 hour mark (infusion completion)
  Compare the impact of a perioperative infusion of oxytocin on perioperative opioid consumption, by comparing the average in perioperative opioids (OMEs)
POD1 Opioid consumption | In the first 24 hours after surgery
  Compare the impact of a perioperative infusion of oxytocin on perioperative opioid consumption, by comparing the average in perioperative opioids (OMEs)
POD2 Opioid consumption | From 24-48 hours after surgery
  Compare the impact of a perioperative infusion of oxytocin on perioperative opioid consumption, by comparing the average in perioperative opioids (OMEs)
POD3 Opioid consumption | From 48-72 hours after surgery
  Compare the impact of a perioperative infusion of oxytocin on perioperative opioid consumption, by comparing the average in perioperative opioids (OMEs)
PACU satisfaction scores | Between 2-4 hours after surgery completion (in the PACU)
  Compare patient postoperative satisfaction scores on an 11 -point Numerical Rating Scale (with 0 being no pain and 10 being worst pain imaginable) between groups
POD1 satisfaction scores | On Post-operative day 1
  Compare patient postoperative satisfaction scores on an 11 -point Numerical Rating Scale (with 0 being no pain and 10 being worst pain imaginable) between groups
POD2 satisfaction scores | On Post-operative day 2
  Compare patient postoperative satisfaction scores on an 11 -point Numerical Rating Scale (with 0 being no pain and 10 being worst pain imaginable) between groups
POD3 satisfaction scores | On Post-operative day 3
  Compare patient postoperative satisfaction scores on an 11 -point Numerical Rating Scale between groups
PACU Post-operative pain | Between 2-4 hours after surgery completion (in the PACU)
  Compare average patient pain scores measured as a mean Brief Pain Inventory (an 11 -point Numerical Rating Scale (with 0 being no pain and 10 being worst pain imaginable)) in PACU after laparoscopic hysterectomy in treated and untreated groups
POD1 Post-operative pain | On Post-operative day 1
  Compare average patient pain scores measured as a mean Brief Pain Inventory (an 11 -point Numerical Rating Scale (with 0 being no pain and 10 being worst pain imaginable)) on POD1 in treated and untreated groups
POD2 Post-operative pain | On Post-operative day 2
  Compare average patient pain scores measured as a mean Brief Pain Inventory (an 11 -point Numerical Rating Scale (with 0 being no pain and 10 being worst pain imaginable)) on POD2 in treated and untreated groups
POD3 Post-operative pain | On Post-operative day 3
  Compare average patient pain scores measured as a mean Brief Pain Inventory (an 11 -point Numerical Rating Scale (with 0 being no pain and 10 being worst pain imaginable)) on POD3 in treated and untreated groups
Intraoperative hypotension (# of episodes of MAP <60 mmHg) | Through surgery completion, an average of 2 hours (From start of infusion to completion end of time in the operating room)
  Assess the impact of a perioperative infusion of oxytocin on hypotension
PACU hypotension (# of episodes of MAP <60 mmHg) | Between 0-4 hours after surgery completion (in the PACU)
  Assess the impact of a perioperative infusion of oxytocin on hypotension

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soffin EM, Lee BH, Kumar KK, Wu CL. The prescription opioid crisis: role of the anaesthesiologist in reducing opioid use and misuse. Br J Anaesth. 2019 Jun;122(6):e198-e208. doi: 10.1016/j.bja.2018.11.019. Epub 2018 Dec 28. PMID 30915988
- [Background] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Background] Bae S, Alboog A, Esquivel KS, Abbasi A, Zhou J, Chui J. Efficacy of perioperative pharmacological and regional pain interventions in adult spine surgery: a network meta-analysis and systematic review of randomised controlled trials. Br J Anaesth. 2022 Jan;128(1):98-117. doi: 10.1016/j.bja.2021.08.034. Epub 2021 Nov 10. PMID 34774296
- [Background] Lundeberg T, Uvnas-Moberg K, Agren G, Bruzelius G. Anti-nociceptive effects of oxytocin in rats and mice. Neurosci Lett. 1994 Mar 28;170(1):153-7. doi: 10.1016/0304-3940(94)90262-3. PMID 8041495
- [Background] Biurrun Manresa JA, Schliessbach J, Vuilleumier PH, Muller M, Musshoff F, Stamer U, Stuber F, Arendt-Nielsen L, Curatolo M. Anti-nociceptive effects of oxytocin receptor modulation in healthy volunteers-A randomized, double-blinded, placebo-controlled study. Eur J Pain. 2021 Sep;25(8):1723-1738. doi: 10.1002/ejp.1781. Epub 2021 May 3. PMID 33884702
- [Background] Matsuura T, Motojima Y, Kawasaki M, Ohnishi H, Sakai A, Ueta Y. [Relationship Between Oxytocin and Pain Modulation and Inflammation]. J UOEH. 2016;38(4):325-334. doi: 10.7888/juoeh.38.325. Japanese. PMID 27980316
- [Background] Gimpl G, Fahrenholz F. The oxytocin receptor system: structure, function, and regulation. Physiol Rev. 2001 Apr;81(2):629-83. doi: 10.1152/physrev.2001.81.2.629. PMID 11274341
- [Background] Baribeau DA, Anagnostou E. Oxytocin and vasopressin: linking pituitary neuropeptides and their receptors to social neurocircuits. Front Neurosci. 2015 Sep 24;9:335. doi: 10.3389/fnins.2015.00335. eCollection 2015. PMID 26441508
- [Background] Miranda-Cardenas Y, Rojas-Piloni G, Martinez-Lorenzana G, Rodriguez-Jimenez J, Lopez-Hidalgo M, Freund-Mercier MJ, Condes-Lara M. Oxytocin and electrical stimulation of the paraventricular hypothalamic nucleus produce antinociceptive effects that are reversed by an oxytocin antagonist. Pain. 2006 May;122(1-2):182-9. doi: 10.1016/j.pain.2006.01.029. Epub 2006 Mar 9. PMID 16527400
- [Background] Yang J. Intrathecal administration of oxytocin induces analgesia in low back pain involving the endogenous opiate peptide system. Spine (Phila Pa 1976). 1994 Apr 15;19(8):867-71. doi: 10.1097/00007632-199404150-00001. PMID 8009342
- [Background] Madrazo I, Franco-Bourland RE, Leon-Meza VM, Mena I. Intraventricular somatostatin-14, arginine vasopressin, and oxytocin: analgesic effect in a patient with intractable cancer pain. Appl Neurophysiol. 1987;50(1-6):427-31. doi: 10.1159/000100753. PMID 2897190
- [Background] Ende HB, Soens MA, Nandi M, Strichartz GR, Schreiber KL. Association of Interindividual Variation in Plasma Oxytocin With Postcesarean Incisional Pain. Anesth Analg. 2019 Oct;129(4):e118-e121. doi: 10.1213/ANE.0000000000003567. PMID 29916862
- [Background] ACOG Practice Bulletin No. 107: Induction of labor. Obstet Gynecol. 2009 Aug;114(2 Pt 1):386-397. doi: 10.1097/AOG.0b013e3181b48ef5. No abstract available. PMID 19623003
- [Background] Kovacheva VP, Soens MA, Tsen LC. A Randomized, Double-blinded Trial of a "Rule of Threes" Algorithm versus Continuous Infusion of Oxytocin during Elective Cesarean Delivery. Anesthesiology. 2015 Jul;123(1):92-100. doi: 10.1097/ALN.0000000000000682. PMID 25909969
- [Background] Heesen M, Carvalho B, Carvalho JCA, Duvekot JJ, Dyer RA, Lucas DN, McDonnell N, Orbach-Zinger S, Kinsella SM. International consensus statement on the use of uterotonic agents during caesarean section. Anaesthesia. 2019 Oct;74(10):1305-1319. doi: 10.1111/anae.14757. Epub 2019 Jul 25. PMID 31347151